CLINICAL TRIAL: NCT02715466
Title: Prospective, Controlled, Double-Blind, Randomized Multicentric Study On The Efficacy And Safety Of An Early Target Controlled Plasma Volume Replacement Therapy With A Balanced Gelatine Solution vs A Balanced Electrolyte Solution In Patients With Severe Sepsis
Brief Title: Gelatin in ICU and Sepsis
Acronym: GENIUS
Status: Terminated | Phase: Phase 4 | Type: Interventional
Why Stopped: recommended by DSMB
Sponsor: B. Braun Melsungen AG (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: HC-G-H-1209
Record Dates: First submitted 2016-03-17; First posted 2016-03-22 (Estimated); Results first posted 2025-08-19 (Actual); Last update posted 2025-08-19 (Actual); Status verified 2025-08

CONDITIONS: Hypovolemia
MeSH Terms: conditions — Hypovolemia

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Gelatine (Experimental): Balanced gelatine solution
  Interventions: Drug: Balanced gelatine solution; Drug: Balanced electrolyte solution
- Electrolyte (Active Comparator): Balanced electrolyte solution
  Interventions: Drug: Balanced electrolyte solution

INTERVENTIONS:
Drug: Balanced gelatine solution — Gelaspan combined with Sterofundin ISO
  Arms: Gelatine
Drug: Balanced electrolyte solution — Sterofundin ISO

SUMMARY:
This prospective, double-blind randomized controlled trial evaluates the differences in terms of efficacy and safety of gelatin based resuscitation as compared to crystalloid based resuscitation in two parallel groups of patients with severe sepsis / septic shock.

ELIGIBILITY:
Inclusion Criteria:

* Male or female patients ≥ 18 years of age
* Women of child bearing potential must test negative on standard pregnancy test (urine or serum)
* Patients with body weight ≤ 140 kg
* Patients diagnosed severe sepsis / septic shock at admission on Intensive Care Unit who can be enrolled within 90 min after admission OR patients diagnosed severe sepsis / septic shock during Intensive Care Unit stay who can be enrolled within 90 min after diagnosis
* Patients where antibiotic therapy has already been started (prior to randomization)
* Patient who are fluid responsive. Fluid responsiveness is defined as increase of > 10% in mean arterial pressure (MAP) after passive leg raising (PLR)
* Signed informed consent by patient, legal representative or authorized person or deferred consent

Exclusion Criteria:

* Administration of HES, dextrane solutions or > 500 ml of Gelatin solutions within the 24 h prior to randomization
* Death expected within the next 48 h (moribund patients as defined by ASA ≥ class V)
* Patients for whom the need of pressure infusions are expected
* Patients with confirmed acute SARS-CoV-2 (COVID-19) infection (as available from routine medical records/ patient chart)
* Requirement for renal support (either continuous or discontinuous techniques, including intermittent haemodialysis, haemofiltration and haemodiafiltration)
* Patients receiving therapeutic heparin medication due to chronic coagulation disease / anticoagulation medication (i.e. partial thromboplastin time > 60 sec)
* Acutely burned patients
* Contraindications according to summary of product characteristics of investigational test and reference product
* Simultaneous participation in another interventional clinical trial (drugs or medical devices studies)

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 167 (Actual)
Dates: Start 2016-04; Primary Completion 2021-12-08 (Actual); Study Completion 2021-12-08 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Gernot Marx, Prof. Dr. med., Study Chair — Universitätsklinikum Aachen,Klinik für Operative Intensivmedizin
Locations (12):
- Medizinische Universität Innsbruck, Innsbruck, Austria
- Masarykova nemocnice v Ústí nad Labem, o.z., Ústí nad Labem, Czechia
- France (2):
  - Université de Nantes, Nantes
  - Hôpital Pasteur 2 - CHU de Nice, Nice
- Germany (6):
  - Universitätsklinikum Aachen, Aachen
  - Klinikum Bremen-Mitte, Bremen
  - Universitätsklinikum Frankfurt, Frankfurt am Main
  - Universitätsinstitut - Johannes Wesling Klinikum Minden, Minden
  - Universitätsmedizin Rostock, Rostock
  - Universitätsklinikum Tübingen, Tübingen
- Spain (2):
  - Hospital Universitari Vall d'Hebron, Barcelona
  - Hospital Universitario La Paz, Madrid

REFERENCES:
- [Derived] Marx G, Zacharowski K, Ichai C, Asehnoune K, Cerny V, Dembinski R, Ferrer Roca R, Fries D, Molnar Z, Rosenberger P, Sanchez-Sanchez M, Schurholz T, Dehnhardt T, Schmier S, von Kleist E, Brauer U, Simon TP. Efficacy and safety of early target-controlled plasma volume replacement with a balanced gelatine solution versus a balanced electrolyte solution in patients with severe sepsis/septic shock: study protocol, design, and rationale of a prospective, randomized, controlled, double-blind, multicentric, international clinical trial : GENIUS-Gelatine use in ICU and sepsis. Trials. 2021 Jun 2;22(1):376. doi: 10.1186/s13063-021-05311-8. PMID 34078421

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Gelatine | Electrolyte
Started | 83 | 84
Completed | 83 | 84
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Gelatine | Electrolyte | Total
Number analyzed (Participants) | 83 | 84 | 167
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 29 | 34 | 63
  >=65 years | 54 | 50 | 104
Age, Continuous [Mean (Standard Deviation); unit: years] | 65.3 (14.20) | 65.9 (14.14) | 65.6 (14.13)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 21 | 20 | 41
  Male | 62 | 64 | 126
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 0 | 0 | 0
  White | 82 | 83 | 165
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 1 | 1 | 2
Region of Enrollment [Number; unit: participants]
  Austria | 6 | 6 | 12
  Czechia | 10 | 9 | 19
  France | 0 | 2 | 2
  Germany | 59 | 61 | 120
  Spain | 8 | 6 | 14

OUTCOME MEASURES:

1. Primary Outcome: Time Until First/Initial Hemodynamic Stabilization
Description: Time from first administration of IMP to first achievement of confirmed hemodynamic stability
Time Frame: 48 hours after treatment start
Population: Intent-to-treat set
Measure: Mean (Standard Deviation); unit: hours
Arm/Group | Gelatine | Electrolyte
Number analyzed (Participants) | 77 | 74
hours | 4.7 (5.88) | 5.8 (6.46)

2. Secondary Outcome: Length of Stay (LOS) in the Intensive Care Unit (ICU)
Description: Length of stay (LOS) in the intensive care unit (ICU)= Date of ICU discharge - date of ICU admission + 1
Time Frame: Intensive care unit (ICU) discharge or day 28
Population: Intent-to-treat set
Measure: Mean (Standard Deviation); unit: days
Arm/Group | Gelatine | Electrolyte
Number analyzed (Participants) | 55 | 53
days | 11.9 (9.32) | 12.8 (10.98)

ADVERSE EVENTS:
Time Frame: From randomization until ICU discharge or day 28- whatever occurs first (max. 28 days)
Arm/Group | Gelatine | Electrolyte
All-Cause Mortality (participants affected / at risk) | 11/83 | 18/84
Serious Adverse Events (participants affected / at risk) | 30/83 | 34/84
Other Adverse Events (participants affected / at risk) | 55/83 | 54/84
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Gelatine (N=83) | Electrolyte (N=84)
Septic shock (Infections and infestations) | 6 (6) | 9 (9)
Abdominal abscess (Infections and infestations) | 0 (0) | 2 (2)
Pneumonia (Infections and infestations) | 2 (2) | 0 (0)
Abscess neck (Infections and infestations) | 0 (0) | 1 (1)
Necrotising fasciitis (Infections and infestations) | 1 (1) | 0 (0)
Pulmonary sepsis (Infections and infestations) | 1 (1) | 0
Multiple organ dysfunction syndrome (General disorders) | 7 (7) | 12 (12)
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 4 (4)
Acute respiratory distress syndrome (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 1 (1)
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 1 (1)
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 1 (1)
Acute respiratory failure (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Bronchial obstruction (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Haemothorax (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Obstructive airways disorder (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Cardiac arrest (Cardiac disorders) | 0 (0) | 4 (5)
Atrial fibrillation (Cardiac disorders) | 2 (2) | 1 (1)
Ventricular tachycardia (Cardiac disorders) | 0 (0) | 3 (3)
Acute myocardial infarction (Cardiac disorders) | 1 (1) | 0 (0)
Bradycardia (Cardiac disorders) | 0 (0) | 1 (1)
Cardiac failure (Cardiac disorders) | 1 (1) | 0 (0)
Pericardial effusion (Cardiac disorders) | 0 (0) | 1 (1)
Right ventricular failure (Cardiac disorders) | 1 (1) | 0 (0)
Tachyarrhythmia (Cardiac disorders) | 1 (1) | 0 (0)
Failure to anastomose (Injury, poisoning and procedural complications) | 3 (3) | 3 (3)
Gastrointestinal anastomotic leak (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Postoperative delirium (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Subdural haematoma (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Suture rupture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Transfusion reaction (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Weaning failure (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Intestinal ischaemia (Gastrointestinal disorders) | 2 (2) | 1 (1)
Duodenal perforation (Gastrointestinal disorders) | 0 (0) | 1 (1)
Duodenal stenosis (Gastrointestinal disorders) | 0 (0) | 1 (1)
Gastric perforation (Gastrointestinal disorders) | 0 (0) | 1 (1)
Ileus (Gastrointestinal disorders) | 0 (0) | 1 (1)
Ileus paralytic (Gastrointestinal disorders) | 1 (1) | 0 (0)
Intestinal haemorrhage (Gastrointestinal disorders) | 1 (1) | 0 (0)
Intra-abdominal haematoma (Gastrointestinal disorders) | 0 (0) | 1 (1)
Pancreatitis acute (Gastrointestinal disorders) | 1 (1) | 0 (0)
Hypotension (Vascular disorders) | 2 (2) | 2 (2)
Haemorrhage (Vascular disorders) | 1 (1) | 1 (1)
Circulatory collapse (Vascular disorders) | 0 (0) | 1 (1)
Shock haemorrhagic (Vascular disorders) | 1 (1) | 1 (1)
Haematoma (Vascular disorders) | 1 (1) | 0 (0)
Haemodynamic instability (Vascular disorders) | 0 (0) | 1 (1)
Hypovolaemic shock (Vascular disorders) | 1 (1) | 0 (0)
Ischaemia (Vascular disorders) | 1 (1) | 0 (0)
Brain injury (Nervous system disorders) | 0 (0) | 2 (2)
Cerebral infarction (Nervous system disorders) | 1 (1) | 1 (1)
Cerebral haematoma (Nervous system disorders) | 1 (1) | 0 (0)
Epilepsy (Nervous system disorders) | 0 (0) | 1 (1)
Generalised tonic-clonic (Nervous system disorders) | 0 (0) | 1 (1)
Paraplegia (Nervous system disorders) | 1 (1) | 0 (0)
Seizure (Nervous system disorders) | 0 (0) | 1 (1)
Somnolence (Nervous system disorders) | 1 (1) | 0 (0)
Spinal cord ischaemia (Nervous system disorders) | 1 (1) | 0 (0)
Antiphospholipid syndrome (Blood and lymphatic system disorders) | 1 (1) | 0 (0)
Coagulopathy (Blood and lymphatic system disorders) | 0 (0) | 1 (1)
Splenic infarction (Blood and lymphatic system disorders) | 0 (0) | 1 (1)
Hepatic failure (Hepatobiliary disorders) | 1 (1) | 1 (1)
Hepatic infarction (Hepatobiliary disorders) | 0 (0) | 1 (1)
Acute kidney injury (Renal and urinary disorders) | 2 (2) | 1 (1)
Explorative laparotomy (Surgical and medical procedures) | 0 (0) | 1 (1)
Leg amputation (Surgical and medical procedures) | 1 (1) | 0 (0)
Hypoglycaemia (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
Device occlusion (Product Issues) | 1 (1) | 0 (0)
Brain Oedema (Nervous system disorders) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 4% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Gelatine (N=83) | Electrolyte (N=84)
Hypernatraemia (Metabolism and nutrition disorders) | 9 (9) | 5 (5)
Iron deficiency (Metabolism and nutrition disorders) | 0 (0) | 4 (4)
Hypoalbuminaemia (Metabolism and nutrition disorders) | 3 (3) | 4 (4)
Hypokalaemia (Metabolism and nutrition disorders) | 2 (2) | 5 (5)
Hyperglycaemia (Metabolism and nutrition disorders) | 2 (2) | 4 (4)
Hypocalcaemia (Metabolism and nutrition disorders) | 4 (4) | 1 (1)
Anaemia (Blood and lymphatic system disorders) | 15 (15) | 15 (16)
Thrombocytosis (Blood and lymphatic system disorders) | 4 (4) | 10 (10)
Thrombocytopenia (Blood and lymphatic system disorders) | 6 (6) | 4 (4)
Atrial fibrillation (Cardiac disorders) | 9 (9) | 10 (12)
Bradycardia (Cardiac disorders) | 4 (4) | 2 (2)
Pneumonia (Infections and infestations) | 2 (2) | 4 (4)
Septic shock (Infections and infestations) | 4 (4) | 1 (1)
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 7 (7) | 6 (6)
Haemoglobin decreased (Investigations) | 3 (3) | 4 (4)
Acute kidney injury (Renal and urinary disorders) | 10 (12) | 6 (6)
Intensive care unit acquired weakness (Nervous system disorders) | 1 (1) | 4 (7)
Delirium (Nervous system disorders) | 3 (3) | 5 (5)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of 60 days or less

DOCUMENTS (2):
  • Study Protocol (2020-06-16): https://cdn.clinicaltrials.gov/large-docs/66/NCT02715466/Prot_002.pdf
  • Statistical Analysis Plan (2022-07-05): https://cdn.clinicaltrials.gov/large-docs/66/NCT02715466/SAP_001.pdf